CLINICAL TRIAL: NCT04247789
Title: The Fatigue in Older Adults Living in a Rest Home: Prevalence and Associated Factors
Brief Title: The Associated Factors With Fatigue in Older Adults Living in a Rest Home
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Sevim ACARÖZ CANDAN, Phsiotherapy and Rehabilitation Department, Ordu University
Other Study IDs: OrduU7
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Fatigue; Older People--Abuse of
Keywords: fatigue; physical function; strength; older adults; nursing homes
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total sample: This group consists of older adults living in a rest home, who are proper for inclusion criteria
  Interventions: Other: Self-reported questionairres

INTERVENTIONS:
Other: Self-reported questionairres — the fatigue will be determined through self reported questionnairres

SUMMARY:
Fatigue is an important and prevalent problem in older adults. The ratio of fatigue may rise in older adults who live in nursing homes/rest homes. In the literature, a few studies investigated the prevalence of fatigue, and there is no study explaining the associated factors. The aim of the present study is to investigate the prevalence of fatigue in rest home residents and to determine the associated variables with fatigue.

ELIGIBILITY:
Inclusion Criteria:

* age older than 65 years
* able to walk with/without walking device
* living at a rest home for at least 12 months
* being voluntary for all assessments

Exclusion Criteria:

* had a cognitive problem (MMSE<24 scores)
* had a neurologic disorder
* had a cancer history
* had uncontrolled cardiopulmonary dysfunction

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The older adults living in a rest home
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Fall Severity Scale (FSS) | 5 minutes
  The FSS is the most frequently used scale among the unidimensional scales which have been developed to assess fatigue. The scale rates the fatigue with nine items, For each item, the patient is asked to grade the fatigue level between 1 and 7, where 1 indicates strong disagreement and 7 indicates strong agreement. A score of 28 or higher generally indicates presence of fatigue.

SECONDARY OUTCOMES:
Strength assessment | 5 minutes
  Quadriceps strength and handgrip strength will be measured by digital dynamometers named as Lafayette and Jamar dynamometers, respectively. Quadriceps strength will be measured in a sitting position with hip and knee flexed 90 degrees. The participants extend the knee and the examiner applies an opposite force to break this position. This test will be performed three times and the maximum value will be recorded in a kilogram. The handgrip strength will be assessed according to the American Society of Hand Therapists. The participants will be asked to squeeze as forcefull as possible the dynamometer. The maximum score of three trials will be recorded in kliograms.
Functional Capacity | 6-10 minutes
  Six-minutes walk test will be used to evaluate the functional capacity or cardiorespiratory fitness. The participants will be walking in a 30-meter corridor for 6-minutes. If necessary the participants can use the walking assistive devices and take a rest. The total distance will be recorded in meters.
Physical Function | 5 minutes
  Short Physical Performance Battery will be used to measure physical functioning. This battery includes 3 subdomains (gait speed, balance and chair stand test). The totatl score changes between 0 and 12. The higher score indicates better performance.
Boddy mass index | 2 minutes
  The body measures (weight and height) will be assessed in kilograms and meters. The index will be calculated by dividing body weight by height squared.
Physical activity habits | 1 minutes
  Physical activity habits will be determined with a question" How many times did you exercise for 30 minutes or more with a certain tempo?" This question will be recorded as a dichotomous variable, 1 indicates present physical activity habits (>2 times) and 0 no physical activity habits (<3 times).
Body mass | 30 seconds.
  The weight will be measured in kilograms without shoes and within thin clothes
Body Height | 30 seconds
  The height will be determined in an erect standing position as centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Sevim ACARÖZ CANDAN, Ordu, Altinordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No